CLINICAL TRIAL: NCT03282656
Title: Pilot and Feasibility Study of Hematopoietic Stem Cell Gene Transfer for Sickle Cell Disease
Brief Title: Gene Transfer for Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Williams (Other)
Responsible Party: Sponsor-Investigator, David Williams, Chief Scientific Officer, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00026188
Record Dates: First submitted 2017-08-22; First posted 2017-09-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: Gene therapy; lentivirus vector; BCL11A; Fetal Hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, single center, pilot and feasibility, single arm cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): open-label, non-randomized, single center, pilot and feasibility, single arm cohort study of a single infusion of autologous bone marrow derived CD34+ HSC cells transduced with lentiviral vector containing a short-hairpin RNA targeting BC11A.
  Interventions: Biological: single infusion of autologous bone marrow derived CD34+ HSC cells transduced with the lentiviral vector containing a short-hairpin RNA targeting BCL11a

INTERVENTIONS:
Biological: single infusion of autologous bone marrow derived CD34+ HSC cells transduced with the lentiviral vector containing a short-hairpin RNA targeting BCL11a — single infusion of autologous bone marrow derived CD34+ HSC cells transduced with the lentiviral vector containing a short-hairpin RNA targeting BCL11a

SUMMARY:
A promising approach for the treatment of genetic diseases is called gene therapy. Gene therapy is a relatively new field of medicine that uses genetic material (mostly DNA) from the patient to treat his or her own disease. In gene therapy, the investigators introduce new genetic material in order to fix or replace the patient's disease gene, with the goal of curing the disease. The procedure is similar to a bone marrow transplant, in that the patient's malfunctioning blood stem cells are reduced or eliminated using chemotherapy, but it is different because instead of using a different person's (donor) blood stem cells for the transplant, the patient's own blood stem cells are given back after the new genetic material has been introduced into those cells. This approach has the advantage of eliminating any risk of GVHD, reducing the risk of graft rejection, and may also allow less chemotherapy to be utilized for the conditioning portion of the transplant procedure. The method used to introduce the gene into the patient's own blood stem cells is to engineer and use a modified version of a virus (called a 'vector') that efficiently inserts the "correcting" genetic material into the cells. The vector is a specialized biological medicine that has been formulated for use in human beings.

The investigators have recently discovered a gene that is very important in the control of fetal hemoglobin expression. Increasing the expression of this gene in sickle cell patients could increase the amount of fetal hemoglobin while simultaneously reducing the amount of sickle hemoglobin in their blood, and therefore potentially cure the condition. In summary, the advantages of a gene therapy approach include: 1) it can be used even if the patient does not have a matched donor available; 2) it may allow a reduction in the amount of chemotherapy required to prepare the patient for the transplant; and 3) it will avoid the strong medicines often required to prevent and treat GVHD and rejection. The goal is to test whether this approach is safe, and whether using gene therapy to change the expression of this particular gene will lead to increased fetal hemoglobin production in people with sickle cell disease.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, single center, pilot and feasibility, single arm cohort study involving a single infusion of autologous bone marrow derived CD34+ HSC cells transduced with the lentiviral vector containing a short-hairpin RNA targeting BCL11a. Accrual will be a maximum of 7 evaluable patients with SCD. The study will have three strata:

1. Stratum 1: ages ≥18-40
2. Stratum 2: ages ≥12-<18
3. Stratum 3: ages ≥3-<12

To determine the feasibility and safety of administering a lentiviral gene transfer vector encoding a small hairpin (sh) RNA targeting the γ-globin gene repressor, BCL11A, in patients with severe SCD.

Patients will undergo standard work-up for autologous bone marrow transplantation according to institutional guidelines and then undergo two bone marrow harvests at a minimum of 4 weeks apart that will be used for a back-up marrow (minimum of 2 x 106 CD34+ cells/kg) and for a harvest of autologous bone marrow for gene transfer.

Patients will receive blood transfusions for a period of 3 months prior to the planned date of product infusion, with a goal of achieving a HbS level ≤ 30% by the time of gene transfer. If the subject is already on a chronic transfusion regimen as part of baseline disease management, the regimen may be continued. The timing of transfusions will be coordinated to occur within 7 days prior to any procedures requiring anesthesia such as bone marrow harvest.

Hematopoietic cells will be collected from the patient in advance of the treatment, to serve as a salvage procedure ("back-up graft"), should there be no hematopoietic recovery observed following the injection of genetically-manipulated cells, or should manipulated cells fail to meet release criteria. Bone marrow (up to 20 mL/kg) will be harvested from the patient under general anesthesia from the posterior iliac crests on both sides by multiple punctures at a minimum of 4 weeks prior to gene therapy. A portion of the bone marrow containing at least 2 x 106 CD34+ cells/kg will be frozen and stored unmanipulated according to standard clinical procedures for autologous bone marrow collection to constitute the back-up graft. If the number of CD34+ cells that exceeds 2 x 106 cells/kg is greater than or equal to 1 x 106 cells/kg, these excess cells would be processed for transduction, transduced, and then frozen. Transduction will be carried out on the selected CD34+ cells and transduced cells will be cryopreserved. If cells from the first harvest were transduced and frozen, these gene-modified cells will be thawed and prepared for infusion in parallel with the product from the subsequent harvest(s). In this case two separate products would be infused. All cell manipulation procedures and release testing will be performed in the transduction facility in accordance with Good Manufacturing Practice (GMP) following process specific standard operating procedures. Final Drug Product will be accompanied by a Certificate of Analysis, documenting that all release testing is complete and within specification. Subjects will receive myeloablative conditioning with Busulfan administered on days -5 to -2, prior to infusion of transduced cells. Cells will be infused intravenously over 30-45 minutes after standard prehydration and premedication according to Boston Children's Hospital Hematopoietic Stem Cell Transplantation Unit standard guidelines. This standard requires that the patient be on continuous cardiac, respiratory and oxygen saturation monitor throughout the infusion and for 30 minutes afterwards. Vital signs will be measured and recorded pre-transfusion, 15 minutes into transfusion, every hour for duration of infusion, and end of transfusion. The RN will stay with the patient for the first 5 minutes of the transfusion. If two transduction products are administered, the second transduced product will be administered without delay after the first.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD with genotype HbSS, HbS/0 thalassemia, HbSD, or HbSO
* Severe symptomatic SCD, defined by the presence of one or more of the following clinical complications:

  1. Minimum of two episodes of acute chest syndrome (ACS) in the 2 years before study entry.
  2. History of three or more episodes of severe pain events requiring a visit to a medical facility and treatment with parenteral opioids in the 2 years before study entry.
  3. Recurrent priapism (> 2 episodes) in the 2 years before study entry.
  4. Red-cell alloimmunization (>2 antibodies) during long-term transfusion therapy.
  5. Receiving, or indicated to receive (based on prior stroke or elevated transcranial Doppler (TCD) results), chronic transfusions for primary or secondary stroke prophylaxis.
* Age 3 years to 40 years .
* Failure of hydroxyurea therapy due to lack of clinical improvement or inability to tolerate due to side effects (e.g., myelosuppression, gastrointestinal symptoms, or hepatic enzyme elevations). Clinical criteria must be met despite taking hydroxyurea for greater than or equal to 6 months, unless contraindicated or not tolerated. Patients taking hydroxyurea who still meet all inclusion criteria are eligible for the trial.
* No HLA-genotypically identical related bone marrow donor available
* Parental/guardian/patient signed informed consent
* Willingness to return for follow-up for 15 years
* White blood cell (WBC) count within the range of 3.0 - 20.0 x 109 /L Hemoglobin within the range of 5 - 11 g/dL Platelet count within the range of 100 - 600 x 109 /L PT and PTT within normal limits, unless prolonged due to anticoagulation requirement.
* Adequate organ function and performance status:

  1. Performance status ≥70% (Lansky play for age <16 years, Karnofsky for age ≥16 years)
  2. Left ventricular ejection fraction >40% or shortening fraction >25%
  3. Direct bilirubin ≤ 2.0 mg/dL
  4. Serum creatinine </= 1.5 times the upper limit of normal for age, and creatinine clearance or GFR >/= 70 mL/min/1.73 m2.
  5. For ages > 7 years, DLCO (corrected for hemoglobin), FEV1, FVC >50% of predicted; if age < 7 years, then oxygen saturation >92% on room air.

Exclusion Criteria:

* Contraindication to bone marrow harvest, or to administration of conditioning medication (busulfan).
* Subjects who have undergone allogeneic transplant previously.
* Known positive HIV serology or HIV nucleic acid testing, or positive serology for HCV, HBV, or HTLV.
* Uncontrolled infection.
* Active malignancy.
* Known myelodysplasia of the bone marrow or abnormal bone marrow cytogenetics.
* Receipt of an investigational study drug or procedure within 90 days of study enrollment.
* Pregnancy, or breastfeeding in a postpartum female, or absence of adequate contraception for fertile subjects. Females of child-bearing potential must agree to use a medically acceptable method of birth control such as oral contraceptive, intrauterine device, barrier and spermicide, or contraceptive implant/injection from Screening through at least 6 months after drug product infusion. Male subjects must agree to use effective contraception (including condoms) from Screening through at least 6 months after drug product infusion.
* Acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on prior biopsy.
* An assessment by the Investigators that the subject will not comply with the study procedures outlined in the study protocol

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Rescue of hematopoiesis after conditioning | within 7 weeks following infusion of gene transfer product
  Rescue of hematopoiesis after conditioning (defined by absolute neutrophil count (ANC) greater than or equal to 0.5 x 109 /L for three consecutive days), achieved within 7 weeks following infusion (i.e., "primary engraftment").

SECONDARY OUTCOMES:
Expression of transgene | at 6 weeks post gene transfer then every 6 months until 2 years after gene transfer
  a. Presence of the transgene (vector copy number) in the following samples: i) Peripheral blood cells [measured in whole blood, mononuclear cells, and the following sorted populations: CD3+, CD15+, CD19+, and CD56+] at 6 weeks, and then every 6 months until 2 years after gene transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Esrick, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - UCLA - Mattel Children's Hospital, Los Angeles, California
  - Boston Children's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esrick EB, Lehmann LE, Biffi A, Achebe M, Brendel C, Ciuculescu MF, Daley H, MacKinnon B, Morris E, Federico A, Abriss D, Boardman K, Khelladi R, Shaw K, Negre H, Negre O, Nikiforow S, Ritz J, Pai SY, London WB, Dansereau C, Heeney MM, Armant M, Manis JP, Williams DA. Post-Transcriptional Genetic Silencing of BCL11A to Treat Sickle Cell Disease. N Engl J Med. 2021 Jan 21;384(3):205-215. doi: 10.1056/NEJMoa2029392. Epub 2020 Dec 5. PMID 33283990